CLINICAL TRIAL: NCT06598878
Title: Effect of AR Environment Stimulation on Proactive and Reactive Modulation of Gait in Individuals With Parkinson Disease
Brief Title: AR Gait Training for Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD_001
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: PD - Parkinson's Disease
Keywords: Augmented Reality; Gait Taining; Heart Rate Variability (HRV)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients (Experimental): AR gait training
  Interventions: Procedure: AR gait training
- PD patients (Control) (No Intervention): Control Group

INTERVENTIONS:
Procedure: AR gait training — Participants will walk on a pathway projected in augmented reality (AR), following the instructions provided on the pathway Each session will last for 60 minutes, conducted three times per week, over a period of six weeks.
  Arms: PD patients

SUMMARY:
Gait disorders in Parkinson's disease (PD), particularly in complex environments or under stress, present challenges for accurate evaluation and classification, such as in cases of freezing of gait. Traditional clinical and laboratory settings often fail to replicate the complexity needed for precise classification, making effective rehabilitation difficult. This study aims to address these challenges by developing an augmented reality (AR)-based environment that mimics real-world stressors and dynamically adapts to the patient's condition. The AR system is designed to facilitate individualized gait training and rehabilitation by modifying environmental difficulty based on real-time feedback from gait performance and stress levels.

Building on Gentile's taxonomy of tasks, the investigators have incorporated PD-specific factors, such as cognitive dual tasks, into our environment classification system. Preliminary results suggest that this system effectively elicits varying gait and heart rate variability (HRV) responses, indicating different stress levels.

This trial will further test the AR environment's ability to classify patients based on their responses to complex, interactive environments, while also investigating the effects of adaptive AR-based gait training on both gait and stress management in individuals with PD.

DETAILED DESCRIPTION:
Gait disorder in Parkinson's disease (PD), has been reported to be related to complex environments and stress situations. To perform precise evaluation on gait disorder, such as freezing of gait, is not easy in clinical and/or lab environment, causing the difficulty to make accurate classification of gait disorder. Designing a standard environment stimulation paradigm helps to promote precise classification of gait disorders. Monitoring the stress situation that causes gait disorder, and dynamically modifying environment assists in the facilitation of effective individualized gait rehabilitation for PD patients.

Although Gentile's taxonomy of tasks provides a structure to examine the complexity of movement task in accordance with environmental context, this taxonomy and environmental context does not specifically reflects PD movement problems. In this on-going project, the investigators developed an environment classification system based on Gentile's taxonomy, but added PD related factors, such as cognitive dual task to meet the needs of this population. Our preliminary results showed that this novel classification successfully induced different levels of gait and HRV responses, suggesting different stress situations.

For the following, the investigators plan to apply the Augment reality (AR) technique to produce standard interactive testing and training environment. AR allows us to mimic complex environments in lab for evaluation and rehabilitation. In addition, AR could interactively change the difficulty of environment according to the patients'gait and stress situation which is important for developing effective personal rehabilitation program

The purposes for this project are as follows:

1. Test the AR environment stimulation on classifying patients and establish the relationships among challenging AR environment, pressure, and gait
2. Investigate the effects of interactive AR gait training on gait and stress for individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Walking Speed | Baseline, 6 weeks, 8 weeks
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline, 6 weeks, 8 weeks
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Step Time | Baseline, 6 weeks, 8 weeks
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.
Time-Domain Index of Heart Rate Variability (HRV)：Standard deviation of RR intervals (SDRR) | Baseline, 6 weeks, 8 weeks
  SDRR is the standard deviation of all recorded RR intervals (the time between successive heartbeats) over a specific period, usually expressed in milliseconds. This measure captures the total variability in heart rate, representing the physiological responses to a variety of internal and external stimuli. High SDRR values generally indicate greater heart rate variability, which is associated with good cardiovascular health and resilience to stress.
Time-Domain Index of HRV：pNN50 | Baseline, 6 weeks, 8 weeks
  Percentage of successive RR intervals that differ by more than 50 ms. pNN50 reflects beat-to-beat variance in heart rate and is considered an indicator of parasympathetic nervous system activity, specifically linked to vagal tone. A higher pNN50 typically indicates better heart rate variability and healthier autonomic function.
Time-Domain Index of HRV：Root mean square of successive RR interval differences (RMSSD) | Baseline, 6 weeks, 8 weeks
  RMSSD is the square root of the mean of the squares of successive differences between adjacent RR intervals. It emphasizes the high-frequency variations in heart rate that are typically mediated by the parasympathetic nervous system
Frequency-Domain Index of HRV: Low Frequency (LF) | Baseline, 6 weeks, 8 weeks
  The LF component typically represents the power of the HRV spectrum in the frequency range of 0.04 to 0.15 Hz. It is measured in milliseconds squared (ms²) or normalized units and is often interpreted as reflecting both sympathetic and parasympathetic activity,
Frequency-Domain Index of HRV: High Frequency (HF) | Baseline, 6 weeks, 8 weeks
  HF typically covers the frequency range from 0.15 to 0.40 Hz and is associated with the respiratory cycle. HF power is usually measured in milliseconds squared (ms²) or normalized units and is indicative of the modulation of heart rate by the parasympathetic nervous system during breathing.
Frequency-Domain Index of HRV: Ratio of LF to HF Power | Baseline, 6 weeks, 8 weeks
  The ratio of LF (low frequency) to HF power in the HRV spectrum. Since LF can represent both sympathetic and parasympathetic activity, comparing it to HF offers insights into the sympathetic-parasympathetic balance
Total Time to Complete the Time Up and Go test | Baseline, 6 weeks, 8 weeks
  The time, in seconds, it takes for a participant to complete the TUG test from the initial sitting position to returning to the seated position.

SECONDARY OUTCOMES:
Double Support Time | Baseline, 6 weeks, 8 weeks
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline, 6 weeks, 8 weeks
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle
Swing Time | Baseline, 6 weeks, 8 weeks
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
Stance Time | Baseline, 6 weeks, 8 weeks
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline, 6 weeks, 8 weeks
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, expressed as steps per minute.
Total UPDRS-III Score | Baseline, 6 weeks, 8 weeks
  The Unified Parkinson's Disease Rating Scale (UPDRS) Part III, also known as the UPDRS-III or the Motor Examination, is a critical component of the UPDRS used to assess the motor symptoms of Parkinson's disease (PD). To provide a comprehensive assessment of motor function in individuals with Parkinson's disease, covering aspects such as bradykinesia (slowness of movement), rigidity, tremors, and postural instability. The UPDRS-III consists of 14 items, each rated on a scale from 0 (normal) to 4 (severe), with a total possible score range from 0 to 108. Higher scores indicate greater motor impairment.
Total NFOG-Q Score | Baseline, 6 weeks, 8 weeks
  The New Freezing of Gait Questionnaire (NFOG-Q) is a specialized tool designed to quantify the severity and impact of freezing of gait (FOG) episodes in individuals with Parkinson's disease (PD). To assess the presence, severity, and impact of FOG in individuals with Parkinson's disease, focusing on how it affects daily activities and mobility. The scores from Parts 2 and 3 are used to calculate a total score that reflects the overall severity and impact of FOG. This total score can help in gauging the effectiveness of treatments aimed at reducing the severity or frequency of FOG episodes.
Overall PDQ-39 Score | Baseline, 6 weeks, 8 weeks
  To evaluate the quality of life across multiple dimensions affected by Parkinson's disease, including mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. The PDQ-39 consists of 39 items, with each item relating to an aspect of life potentially impacted by PD. Responses to these items are aggregated into eight scales corresponding to the dimensions mentioned above.Each item is scored on a scale from 0 (never) to 4 (always), with the total score for each dimension being converted to a 0-100 scale. A higher score indicates a lower quality of life.
Total HADS Score | Baseline, 6 weeks, 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a validated instrument designed to identify and quantify the severity of anxiety and depression symptoms, particularly focusing on the psychological rather than the somatic aspects to avoid confounding with physical illnesses. To screen for, and evaluate the severity of, anxiety and depression symptoms in a wide range of healthcare settings, especially useful in populations where physical illness might overlap with psychological distress. The scores for each subscale (anxiety and depression) range from 0 to 21. These can be combined to give a total HADS score, which ranges from 0 to 42, with higher scores indicating more severe symptoms.
Overall PSQI Score | Baseline, 6 weeks, 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a comprehensive self-rated questionnaire that assesses sleep quality and disturbances over the past month. To evaluate the quality and patterns of sleep, identifying sleep disorders and quantifying the degree of sleep-related problems. Each component is scored on a scale of 0 to 3, with the total PSQI score ranging from 0 to 21. Higher scores indicate poorer sleep quality.
Non-linear Index of HRV: SD1 | Baseline, 6 weeks, 8 weeks
  SD1 is calculated from the Poincaré plot, where it measures the dispersion of points perpendicular to the line of identity, usually expressed in milliseconds. This dispersion specifically quantifies the short-term variability in heart rate, primarily influenced by the parasympathetic nervous system. SD1 provides insight into the rapid changes in heart rate variability, offering a unique perspective on autonomic nervous system activity that traditional time-domain and frequency-domain measures might not fully capture.
Non-linear Index of HRV: SD2 | Baseline, 6 weeks, 8 weeks
  SD2 is calculated as the standard deviation of points along the line of identity in the Poincaré plot, reflecting long-term heart rate variability, usually expressed in milliseconds. This measure captures broader fluctuations in heart rate that are influenced by both sympathetic and parasympathetic nervous system activities. SD2 provides insights into the overall autonomic balance and the body's ability to adapt to sustained physiological stressors or environmental changes. It is particularly useful in studies investigating chronic stress, cardiovascular health, or the impact of long-term interventions.
Non-linear Index of HRV: Ratio of SD1-to-SD2 | Baseline, 6 weeks, 8 weeks
  The SD1/SD2 ratio is calculated by dividing SD1, which measures short-term variability and is predominantly influenced by parasympathetic activity, by SD2, which measures long-term variability and reflects both sympathetic and parasympathetic influences. This ratio is useful for assessing the autonomic balance or the sympathetic-parasympathetic interaction. A higher SD1/SD2 ratio indicates a dominance of parasympathetic activity relative to sympathetic, suggesting a more "relaxed" autonomic state, whereas a lower ratio indicates a relative dominance of sympathetic activity, which could be associated with stress, reduced cardiac health, or other health risks.
Total Montreal Cognitive Assessment (MoCA) Score | Baseline, 6 weeks, 8 weeks
  The MoCA is a widely used cognitive screening tool that assesses multiple cognitive domains, including attention, memory, executive functions, language, visuospatial abilities, and orientation
Total Mini-Mental State Examination (MMSE) Score | Baseline, 6 weeks, 8 weeks
  The MMSE is a widely used cognitive screening tool designed to assess global cognitive function across several domains, including orientation, registration, attention, calculation, recall, and language

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan